CLINICAL TRIAL: NCT06259942
Title: The Effect of Usıng Heated Intravenous Fluıds wıth Underbody Warmers on Maternal and Neonatal Well-Beıng in Cesarean Sectıon Operatıons
Brief Title: Impact of Active Heating on Maternal and Neonatal Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Dilek Talhaoglu, principal investigator, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Surgery-01
Record Dates: First submitted 2024-01-12; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Hypothermia
MeSH Terms: conditions — Hypothermia | interventions — Control Groups; Population Groups

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Masking Description: women undergoing elective caesarean section
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention 1 group (Experimental): only the group heated throughout surgery with carbon fiber underbody heaters
  Interventions: Other: İntervention 1 group (underbody heater group only); Other: Control Group
- Intervention 2 group (Active Comparator): the group that was both warmed throughout the operation with carbon fiber underbody heaters and given warmed intravenous fluids
  Interventions: Other: İntervention 2 group (group using both underbody heater and heated iv liquid)
- Control group (No Intervention): routine practice of the hospital where the surgery was performed (no heater applied group)

INTERVENTIONS:
Other: İntervention 1 group (underbody heater group only) — Resistive heaters can be set to 38-40°C and are used together with the control unit to which they are connected. In the study, an underbody heater (MEDWARM W 300 IM 190MS branded) system measuring 1900x500x40mm was used. In this study, the underbody heater was set to 38°C for patients. Before use, a surgical drape was placed over it to prevent direct patient contact.
  Other Names: MEDWARM W-300 IM-190MS
  Arms: Intervention 1 group
Other: İntervention 2 group (group using both underbody heater and heated iv liquid) — IV fluids should be warmed to protect patients from unwanted hypothermia during surgery. One liter of saline solution given at room temperature decreases body temperature by 0.25˚C in adults. Therefore, the fluids given to the patient should be heated to 33 40˚C. In the guideline published by the Turkish Anesthesia Society, it is stated that if more than 1000 2000 mL of fluid is to be given to patients, it should be heated at 37°C (TARD, 2013). In this study, both IV fluids were heated between 37 and 39°C and given to the patient and heated with carbon fiber underbody heaters.
  Other Names: MEDWARM W-300 IM-190MS, QW3 Blood and Serum Warmer
  Arms: Intervention 2 group
Other: Control Group — no active heating treatment was applied in this group
  Other Names: group without active heating
  Arms: Intervention 1 group

SUMMARY:
This study was conducted to determine the effects of actively warming the patient and using warmed intravenous (IV) fluid during cesarean section on maternal and infant well-being

DETAILED DESCRIPTION:
This study was conducted to determine the effects of actively warming the patient and using warmed intravenous (IV) fluid during cesarean section on maternal and infant well-being.

The study was conducted in a university hospital with a total of 105 women who gave birth by cesarean section randomly selected from 35 intervention 1 (only underbody heater group), 35 intervention 2 (both underbody heater and heated IV fluid group) and 35 control group. The research data were collected with the Individual Information Form, Patient Follow-up Form and Visual Analog Scale. APGAR score, body temperature, cortisol and glucose levels were evaluated in the infant and body temperature, intraoperative bleeding, shivering, postoperative pain, gas and urination were evaluated in the mother between the three groups.

Descriptive statistics, Chi-square, Shapiro Wilks, Friedman, Wilxocon, Kuruskal Wallis and Mann Whitney U test were used in the evaluation of the data and significance level p<0.05 was accepted.

ELIGIBILITY:
Inclusion Criteria:

* Elective cesarean section with spinal anesthesia,
* 37 weeks of gestation and above,
* with ASA I and ASA II scores,
* Pregnant women with a healthy fetus,
* The preoperative fasting period is between 2 to 12 hours,
* Pregnant women who were normothermic (36 to 37.5°C) preoperatively

Exclusion Criteria:

* Those requiring emergency delivery or with comorbidities
* Multiple pregnancies,
* Anemic pregnant women with a hemoglobin value below 11 g/dl according to the World Health Organization (2001),
* Central body temperature above 37.5°C and below 36°C on the morning of surgery
* Pregnant women with a history of malnutrition, thyroid function and other endocrine disorders, Parkinson's disease, peripheral circulatory disorders, diabetes mellitus, heart disease and stroke,
* Pregnant women with chronic bowel problems and urinary system problems were not included in the study.

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 105 (Actual)
Dates: Start 2022-06-19 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Maternal well- being | two day
  body temperature( degrees cantigrade), intraoperative bleeding (hemoglobin) , shivering(0-10) , postoperative pain (0-10), gas and urination

SECONDARY OUTCOMES:
Newborn well- being | two day
  body tempereture (degrees cantigrade), APGAR score , cortisol and glucose levels

CONTACTS AND LOCATIONS:
Overall Officials: Dilek TALHAOĞLU, PhD, Principal Investigator — She was a doctoral student at Erciyes University, Institute of Health Sciences.
Locations (1):
- Erciyes Unıversty, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
December 2025